CLINICAL TRIAL: NCT04684498
Title: An Open-label Study to Evaluate the Efficacy of Neuraminidase Inhibitor Treatment in ST-Elevation Myocardial Infarction (STEMI) Patients
Brief Title: Open-label Study of Neuraminidase Inhibitor Treatment in STEMI Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Dao Wen Wang, Prof., Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-AMI-NI
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: ST Elevation Myocardial Infarction; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamiflu (Oseltamivir Phosphate Capsules) (Experimental): Standardized STEMI treatment + oseltamivir phosphate capsule (75mg, 2 times/day, 7days, oral)
  Interventions: Drug: Oseltamivir phosphate capsules
- no intervention (Other): Standardized STEMI treatment + no intervention
  Interventions: Drug: Oseltamivir phosphate capsules

INTERVENTIONS:
Drug: Oseltamivir phosphate capsules — Treatment group vs. Control group
  Other Names: Tamiflu

SUMMARY:
Neuraminidase-1 can cause the removal of terminal sialic acid residues from the cell surface or serum sialyloconjugates. The level of Neu5Ac was positively related to the activity of neuraminidase-1. Elevation of Neu5Ac was observed in myocardial ischemia animal model, as well as patients with coronary artery disease. It is interesting to note that Neu5Ac and its regulatory enzyme neuraminidase-1 seem to play a key role in triggering myocardial ischemic injury. Oseltamivir, a structural mimic of sialic acid, was widely used as anti-influenza drug. It suppressed neuraminidase-1 activity in the heart. Targeting neuraminidase-1 may represent a new therapeutic intervention for coronary artery disease. This project seeks to identify whether neuraminidase inhibitor (Oseltamivir) treatment could decrease the myocardial infarct size in STEMI patients and improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 75, regardless of gender;
2. STEMI should be diagnosed by two attending physicians or above, including history, clinical symptoms and signs;
3. Participate voluntarily and sign informed consent, and can be followed up for more than one month.

Exclusion Criteria:

1. Allergic to oseltamivir;
2. Creatinine clearance rate less than 60%;
3. Severe liver insufficiency;
4. Female patients who have or plan to become pregnant;
5. Life expectancy less than one year;
6. Patients refused to comply with the requirements of this study;
7. According to the discretion of investigator, the patient was unable to complete the study or comply with the requirements of the study (for administrative or other reasons).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial infarct size at 1 week | 1 week
  Myocardial infarct size at 1 week after acute myocardial infarction (quantified by Gadolinium-enhanced MRI).

SECONDARY OUTCOMES:
Myocardial infarct size | 1 week
  Myocardial infarct size under the curve of creatine kinase-MB (CK-MB) and hypersensitive troponin I.
Myocardial infarct size based on culprit vessel with TIMI 0-1 blood flow | 1 week
  Evaluated by coronary angiography and CMR.
The proportion of viable myocardium and ratio of myocardial reperfusion | 1 week
  The proportion of viable myocardium and reperfusion was determined by the range of abnormal enhancement of gadolinium.
Composite end point at 1 week | 1 week
  A composite end point of cardiogenic shock, cardiac death, malignant arrhythmia, and resuscitated cardiac arrest (including ventricular fibrillation) at 1 week.
Myocardial infarct size at 3 month | 3 month
  Myocardial infarct size at 3 month after acute myocardial infarction (quantified by Gadolinium-enhanced MRI).
Composite end point at 6 month | 6 month
  Composite end point at 6 month, including all-cause death, reinfarction, heart failure after myocardial infarction, and rehospitalization of unstable angina at 6 month.

CONTACTS AND LOCATIONS:
Overall Officials: Dao Wen Wang, M.D., Ph.D, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China